CLINICAL TRIAL: NCT01118104
Title: Relationships Between Sickness Absence and Physical, Mental, and Job-related Factors in Patients With Chronic Pulmonary Disease
Brief Title: Sickness Absence Versus Physical, Mental, and Job-related Factors in Patients With Chronic Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GK57
Record Dates: First submitted 2010-04-27; First posted 2010-05-06 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary vocational rehabilitation (Other)
  Interventions: Other: Vocational pulmonary rehabilitation

INTERVENTIONS:
Other: Vocational pulmonary rehabilitation — Multidisciplinary pulmonary rehabilitation with emphasis on vocational issues

SUMMARY:
People with chronic respiratory disease have shortened work life, their disease is associated with greater work disability and they are at greater risk of being unemployed. Lower employment rates and higher sickness absence is expensive for the community and leads to financial as well as social consequences for the individual.

There is a lack of data on factors that can predict sickness absence and disability in patients with pulmonary disease. We therefore want to study a group of people with COPD and asthma referred to our clinic. The study will investigate relationships between sickness absence and exercise capacity, job-related factors, disease severity, self-efficacy, health related quality of life and subjective health complaints.

ELIGIBILITY:
Inclusion Criteria:

* chronic pulmonary disease
* employed
* periods of sickness absence in the year prior to admittance

Exclusion Criteria:

* lack of ability to complete the rehabilitation program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects absent from work more than 10 days 4 weeks prior to follow-up | 12 months
  The subjects are interviewed after 12 months. Number of days absent from work during 4 weeks prior to the interview are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Morten S Ryg, PhD, Study Director — LHL Helse
Locations (1):
- Glittreklinikken, Hakadal, Akershus, Norway